CLINICAL TRIAL: NCT06072482
Title: A Randomized, Double-blind, Placebo-controlled Phase 4 Clinical Trial to Evaluate the Long-term Safety and Efficacy of Avacopan in Participants With Antineutrophil Cytoplasmic Antibody (ANCA)-Associated Vasculitis
Brief Title: A Study to Evaluate Avacopan in Participants With ANCA-associated Vasculitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20220159; EU CT Number (Other: 2023-503184-42)
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Antineutrophil Cytoplasmic Antibody-associated Vasculitis
Keywords: Avacopan; ANCA-associated Vasculitis; AAV
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — avacopan; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A: Avacopan + Standard of Care (SoC) (Experimental): Avacopan 30 mg twice daily for 5 years + SoC background immunosuppressive therapy.
  Interventions: Drug: Avacopan; Drug: Standard of Care
- Group B: Avacopan/Placebo + SoC (Experimental): Avacopan 30 mg twice daily for 1 year, followed by placebo twice daily for 4 years + SoC background immunosuppressive therapy.
  Interventions: Drug: Avacopan; Drug: Placebo; Drug: Standard of Care
- Group C: Placebo + SoC (Placebo Comparator): Placebo twice daily for 5 years + SoC background immunosuppressive therapy.
  Interventions: Drug: Placebo; Drug: Standard of Care

INTERVENTIONS:
Drug: Avacopan — Administered orally.
  Other Names: CCX168
  Arms: Group A: Avacopan + Standard of Care (SoC); Group B: Avacopan/Placebo + SoC
Drug: Placebo — Administered orally.
  Arms: Group B: Avacopan/Placebo + SoC; Group C: Placebo + SoC
Drug: Standard of Care — All participants will receive SoC background immunosuppressive therapy for induction and maintenance, at the discretion of the Investigator and as supported by current guidelines, product labels and local practices and informed by the individual participant's clinical condition, preferences, and values.

SUMMARY:
The primary objective of this study is to evaluate the long-term safety of avacopan in participants with antineutrophil cytoplasmic antibody (ANCA)-associated vasculitis (AAV).

ELIGIBILITY:
Inclusion Criteria:

* Participants has provided informed consent before initiation of any study-specific activities/procedures.
* Newly diagnosed or relapse of granulomatosis with polyangiitis or microscopic polyangiitis, consistent with Chapel-Hill Consensus Conference definitions (Jennette et al, 2013), where induction treatment with cyclophosphamide or rituximab is needed.
* Age >/= 18 years (or >/= legal age within the country if it is older than 18 years).
* Positive test for anti-positive antiproteinase 3 or antimyeloperoxidase (current or historic) antibodies.
* At least 1 Birmingham Vasculitis Activity Score (BVAS) major item, or at least 3 BVAS nonmajor items, or at least the 2 renal items of proteinuria and hematuria.
* eGFR >/= 15 mL/min/1.73 m^2 (using Chronic Kidney Disease Epidemiology Collaboration equations).

Exclusion Criteria:

* Alveolar hemorrhage requiring invasive pulmonary ventilation support anticipated to last beyond the screening period of the study.
* Any other known multisystem autoimmune disease that may confound study assessments and study conclusions including but not limited to eosinophilic granulomatosis with polyangiitis (GPA [Churg-Strauss]), systemic lupus erythematosus, immunoglobulin (Ig) A vasculitis (Henoch-Schönlein), rheumatoid vasculitis, Sjogren's syndrome, anti-glomerular basement membrane disease, or cryoglobulinemic vasculitis.
* Any other medical condition requiring or expected to require continued use of immunosuppressive therapies, including corticosteroids that may cause confoundment with study assessments and study conclusions.
* Received dialysis or plasma exchange within 16 weeks before Day 1 randomization.
* Have had a kidney transplant.
* Malignancy (except curatively treated nonmelanoma skin cancers, curatively treated cervical carcinoma in situ, or breast ductal carcinoma in situ) within the last 5 years before Day 1 randomization.
* Acute or chronic, active hepatitis B virus or hepatitis C virus, or human immunodeficiency virus infection during screening.
* Any known exposure to a case of active tuberculosis (TB) within the last 12 weeks before Day 1 randomization.
* Positive test for active or latent TB during screening.
* White blood cell count < 3500/µL, neutrophil count < 1500/µL, or lymphocyte count < 500/µl. Note: Complete Blood Count can be repeated once in the screening period at the investigator discretion. In such instances, eligibility will be determined based on the repeat complete blood count.
* Evidence of clinically significant hepatic disease including prior diagnosis of cirrhosis.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase (ALP) >2.0 times the upper limit of normal (ULN).
* Total bilirubin > 1.5 times the ULN. Note: A participant with documented Gilbert's syndrome with total bilirubin < 2 x ULN may be eligible.
* Any of the following within 6 weeks prior to Day 1 randomization: serious infection, infection requiring treatment with intravenous (IV) anti-infective agents, any other infection (including active infection, chronic infection, opportunistic infection, or history of recurrent infection) that in the opinion of the investigator would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion. Oral or vaginal candidiasis and cutaneous or nail fungal infections do not constitute an exclusion.
* Any of the following within 12 weeks prior to Day 1 randomization: myocardial infarction, stroke, unstable angina, symptomatic congestive heart failure requiring prescription medication, any other clinically significant cardiovascular disease that in the opinion of the investigator would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.
* Received cyclophosphamide (CYC) within 12 weeks before signing the informed consent; if on azathioprine (AZA), mycophenolate, or methotrexate (MTX) at the time of screening, these drugs must be withdrawn before receiving CYC. Note: If induction therapy with CYC was started within 1 week before signing the informed consent for the current episode of newly diagnosed or relapse of GPA or microscopic polyangiitis (MPA), the participant may be eligible, provided no CYC was received within 12 weeks before the start of the current induction therapy and if on AZA, mycophenolate, or MTX, these were withdrawn prior to receiving the current induction therapy with CYC.
* Have been taking an oral daily dose of a glucocorticoid of more than 10 mg prednisone equivalent for more than 6 weeks continuously before signing of the informed consent.
* Received RTX or other B-cell depleting therapies within 26 weeks before signing of the informed consent; if on AZA, mycophenolate, or MTX at the time of screening, these drugs must be withdrawn before receiving rituximab (RTX). Note: If induction therapy with RTX was started within 1 week before signing the informed consent for the current episode of newly diagnosed or relapse of GPA or MPA, the participant may be eligible, provided no RTX was received within 26 weeks before the start of the current induction therapy and if on AZA, mycophenolate, or MTX, these were withdrawn prior to receiving the current induction therapy with RTX.
* Received any of the following within 16 weeks before Day 1 randomization:
* antitumor necrosis factor treatment
* abatacept
* alemtuzumab
* IV Ig
* belimumab
* anti interleukin-6 agent (eg, tocilizumab, sarilumab).
* Taking a strong or moderate inducer of the cytochrome P450 3A4 (CYP3A4) enzyme unless the strong or moderate CYP3A4 inducer can be changed to an alternative medicine at least 1 week before Day 1 randomization.
* Received an investigational drug within 30 days or within 5 half-lives (whichever is longer) before Day 1 randomization.
* Previously received avacopan without clinical benefit per the Investigator's opinion or received avacopan within 60 days before Day 1 randomization.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2036-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Up to Month 60
Percentage of Participants Experiencing Adverse Events of Special Interest | Up to Month 60
Percentage of Participants Experiencing Serious Adverse Events | Up to Month 60
Percentage of Participants Experiencing Adverse Events Leading to Withdrawal | Up to Month 60
Percentage of Participants Experiencing Adverse Events Leading to Death | Up to Month 60
Number of Participants Experiencing Clinical Significant Changes from Baseline in Vital Signs Measurements | Up to Month 60
Number of Participants Experiencing Clinical Significant Changes from Baseline in Hematology Assessments | Up to Month 60
Number of Participants Experiencing Clinical Significant Changes from Baseline in Serum Chemistry Assessments | Up to Month 60
Number of Participants Experiencing Clinical Significant Changes from Baseline in Urinalysis Assessments | Up to Month 60

SECONDARY OUTCOMES:
Group A and B Participants who Achieved Remission at Month 12: Time to Relapse in AAV Between Month 12 and Month 60 | Month 12 to Month 60
Group A and B Participants who Achieved Remission at Month 12: Percentage of Participants who Relapse After Achieving Remission at Month 12 | Month 12 to Month 60
Groups A and C: Percentage of Participants who Achieved Sustained Remission at Month 60 | Month 60
Group A and C Participants with Overt Renal Disease at Baseline: Change from Baseline to Month 60 in Estimated Glomerular Filtration Rate (eGFR) | Baseline and Month 60
Groups A and C: Change from Baseline to Month 60 in Short Form 36 Health Survey Version 2 (SF-36 v2) General Health Perception Score | Baseline and Month 60
Groups A and C: Change from Baseline to Month 60 in EuroQoL-5 Dimension 5 Levels (EQ-5D-5L) Visual Analogue Scale (VAS) | Baseline and Month 60
Percentage of Participants who Achieved Remission at Month 6 | Month 6
Groups A and C: Change from Baseline to Month 60 in Vasculitis Damage Index (VDI) | Baseline and Month 60
Groups A and C: Percentage of Participants with Composite Outcome of Initiation of Maintenance Dialysis, Kidney Transplantation, or Death | Up to Month 60
Percentage of Participants With Glucocorticoid Use | Up to Month 60
Percentage of Participants With Immunosuppressant Use | Up to Month 60

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (68):
- United States (54):
  - Orthopedic Physicians Alaska, Anchorage, Alaska
  - Scottsdale Healthcare at Shea - HonorHealth, Scottsdale, Arizona
  - Southwest Kidney Institute, Surprise, Arizona
  - Medvin Clinical Research, Covina, California
  - Palo Alto Medical Foundation Fremont, Fremont, California
  - The Nephrology Group, Fresno, California
  - Providence Medical Foundation, Fullerton, California
  - Medvin Clinical Research, Menifee, California
  - University of California San Francisco- Zuckerburg San Francisco General, San Francisco, California
  - Harbor University of California at Los Angeles Medical Center, Torrance, California
  - University of Colorado, Aurora, Colorado
  - Florida Kidney Physicians, Boca Raton, Florida
  - Malcom Randall Veterans Affairs Medical Center, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - ClinTrial Research Oakwater, Llc, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Lake Cumberland Rheumatology, New Albany, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Dunes Clinical Research LLC, Sioux City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Kidney Michigan Institute, Saginaw, Michigan
  - Revive Research Institute, Sterling Heights, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Renown Rheumatology, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - New York Nephrology Vasculitis and Glomerular Center, Albany, New York
  - Northwell Health, Great Neck, New York
  - Hospital For Special Surgery, New York, New York
  - East Carolina University Brody Outpatient Center, Greenville, North Carolina
  - Brookview Hills Research Associates Llc, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Stat Research, Miamisburg, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny Health Network Cancer Institute at Mellon Pavilion, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Nephrology Associates Inc, East Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Renal Disease Research Institute - Landry Office, Dallas, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Nephrology Associates of Northern Virginia Inc, Fairfax, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Rheumatology and Pulmonary Clinic, Beckley, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Czechia (5):
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Revmatologicky ustav, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
- Hungary (2):
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
- Poland (4):
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - Spzoz Centralny Szpital Kliniczny Umed w Lodzi, Lodz
  - Narodowy Instytut Geriatrii Reumatologii i Rehabilitacji im prof dr hab med Eleonory Reicher, Warsaw
  - Wojskowy Instytut Medyczny - Panstwowy Instytut Badawczy Centralny Szpital Kliniczny Mon, Warsaw
- Romania (3):
  - Spitalul Clinic Sf Maria, Bucuresti, Bucharest
  - Spitalul Clinic Dr Ion Cantacuzino, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj, Cluj-Napoca

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com